CLINICAL TRIAL: NCT03737279
Title: Daily Meditation Program in Women Admitted to the Antepartum Unit: A Randomized Controlled Trial
Brief Title: Daily Meditation Program in Women Admitted to the Antepartum Unit
Acronym: Meditate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Morgen Doty, Principal Investigator, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0810
Record Dates: First submitted 2018-10-23; First posted 2018-11-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy, High Risk; Pregnancy Related
Keywords: Pregnancy; Meditation
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation (Experimental): Intervention Group:
  Routine care plus twice daily mindful meditation
  Interventions: Behavioral: Meditation; Behavioral: Routine Care
- Routine care (Active Comparator): Control Group:
  Routine care which includes ACOG educational pamphlets on day 1, 2 and 3 after randomization
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Meditation — Routine care + twice daily meditation per schedule, to start on the day of randomization
  Arms: Meditation
Behavioral: Routine Care — Routine care including ACOG educational pamphlets:
  * Day 1: "Nutrition in Pregnancy"
  * Day 2: "Heart Health for Women"
  * Day 3: "Exercise after Pregnancy"

SUMMARY:
The purpose of this study is to assess whether a daily mindful meditation program for women admitted to the antepartum floor will decrease maternal state anxiety compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* ≥ 23.0 weeks gestation
* Planned inpatient care for > 3 days from randomization
* Women cared for by UT physicians

Exclusion Criteria:

* Known major lethal fetal anomalies (eg. trisomy 13, trisomy 18, anencephaly, Potter's Syndrome)
* Non-English speaking women
* Planned delivery ≤ 3 days from randomization
* Previous fetal surgery in the current pregnancy (twin twin transfusion syndrome laser ablation, spina bifida repair, etc)
* Women who have practiced a form of meditation in the current pregnancy (including yoga) in the last 4 weeks
* Women who are currently using patient-controlled analgesia (PCA) (eg. sickle cell crisis)
* Admission diagnosis of ecclampsia or HELLP (hemolysis, elevated liver enzymes, low platelets) syndrome
* Diagnosed personality disorder including borderline personality disorder, histrionic personality disorder, schizoid personality disorder, schizotypal personality disorder, schizophrenia
* Diagnosed anxiety, depression, bipolar or other psychiatric illness on medications for these disorders
* Non-reassuring fetal heart tracing on admission
* Intrauterine fetal demise at randomization
* Inability to gain access to phone application

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Maternal state anxiety as assessed by the State Anxiety Scale | 1-3 days
  The State Anxiety Scale Ranges from 20 to 80, with higher scores indicating a higher anxiety level.

SECONDARY OUTCOMES:
Maternal state anxiety as assessed by the State Anxiety Scale | 1 to 11 weeks.
  The State Anxiety Scale score ranges from 20 to 80, with higher scores indicating a higher anxiety level.
Stress as assessed by the Perceived Stress Scale | 3 days to 11 weeks.
  The Perceived Stress Scale score ranges from 0 to 40, with higher scores indicating a higher stress level.
Depression as assessed by the Edinburgh Depression Scale | 3 days to 11 weeks.
  The Edinburgh Depression Scale score ranges from 0 to 30, with higher scores indicating a higher depression level.
Patient satisfaction | 3 days to 11 weeks.
  The Patient satisfaction questionnaire will be scored by a 5-point Likert Scale. Two questions will be asked relating to overall experience with the research trial and overall experience in the hospital. Each of the two questions will be rated with a 5-point Likert, with a total score ranging from 2 to 10 and with higher scores indicating a [better/worse] outcome.
Latency period | At delivery.
  Latency period is defined as time from randomization until delivery
Number of meditation sessions | 11 weeks
  Meditation sessions as reported per patient and documented by phone application.
Duration of meditation sessions | 11 weeks
  Meditation duration as reported per patient and documented by phone application.

CONTACTS AND LOCATIONS:
Overall Officials: Morgen S Doty, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doty MS, Chen HY, Ajishegiri O, Sibai BM, Blackwell SC, Chauhan SP. Daily meditation program for anxiety in individuals admitted to the antepartum unit: a multicenter randomized controlled trial (MEDITATE). Am J Obstet Gynecol MFM. 2022 May;4(3):100562. doi: 10.1016/j.ajogmf.2022.100562. Epub 2022 Jan 12. PMID 35031521